CLINICAL TRIAL: NCT01364220
Title: An Investigator-Sponsored,Double Blind,Placebo-controlled,Randomised,Multi-centre Study to Assess the Effects of Very Early Use of Rosuvastatin in Preventing Recurrence of Ischemic Stroke
Brief Title: The Effects of Very Early Use of Rosuvastatin in Preventing Recurrence of Ischemic Stroke
Acronym: EUREKA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Severance Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Ji Hoe Heo, Ji Hoe Heo, Professor, Department of Neurology, Yonsei University College of Medicine, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3560L00087
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Stroke
Keywords: Additional relevant MeSH terms; Stroke; Cerebral Infarction; Cerebrovascular Disorders; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Magnetic Resonance Imaging; Recurrence
MeSH Terms: conditions — Stroke; Cerebral Infarction; Cerebrovascular Disorders; Recurrence | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin 20mg tablet, once daily, for 14 days
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Placebo tablet, once daily, for 14 days
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20mg tablet, once daily, for 14 days
  Other Names: Crestor 20mg
  Arms: Rosuvastatin
Other: Placebo tablet — Placebo tablet, once daily, for 14 days
  Arms: Placebo

SUMMARY:
It is anticipated that 548 subjects will be recruited from approximately 27 centres in South Korea.

This is an investigator-sponsored, double-blind, placebo-controlled, randomized, multi-centre study to assess the effects of rosuvastatin 20 mg compared to placebo in acute ischemic stroke patients, with the first dose within 18 hours after baseline MRI and continued treatment for 14 days.

Subjects will be male or female, over 20 years, with diagnosis of acute ischemic stroke with baseline MRI, and who are either statin-naïve or untreated with statin for the previous 3 months.

The objective would be to compare the recurrence rate of ischemic stroke by comparing the imaging parameters during 14 days of treatment and clinical improvement as defined by percent improvement based on NIHSS scores measurements at baseline, 5 days and 14 days of treatment.

DETAILED DESCRIPTION:
Statins have action mechanisms that may work nicely in preventing recurrence during acute stage of infarction!

First, statins have antithrombotic effects and lower thrombogenicity. Statins prolong time to arterial thrombosis in endothelial injury model, inhibit P-selectin expression and platelet aggregation, reduce platelet PAR-1 thrombin receptor, and reduce tissue factor levels in plasma, its expression on monocyte surface, and atherosclerotic plaques. Second, statins enhance thrombolysis. They reduce PAI-1, increase t-PA activity and reduce fibrinogen level. Combined treatment of statins and t-PA in rats reduces the infarct size and downregulates expression of tissue factor, ICAM-1, vWF, and MMP-9. In addition, t-PA induced toxicity is reversed by statins.

Third, statins have anti-inflammatory actions that can stabilize and even regress plaques. Statins reduce the number of T-lymphocytes within plaques, inhibit migration and activation of monocyte/macrophage system, and reduce matrix metalloproteinase activity that play a critical role in plaque rupture. Rosuvastatin 40 mg could regress coronary atheroma burden at 2 years, and reduce progression of carotid intima-media thickness.

Benefits of statins in stroke patients are partially proven!

First, statins are well known to be effective in primary prevention of stroke. Second, statins were effective in secondary prevention of stroke. A high dose of statin (atorvastatin 80 mg) reduced recurrent stroke in patients with recent TIA or ischemic stroke when it was administrated 1-6 months after stroke onset. However, it is uncertain whether statins are effective during the first month after stroke. Third, outcomes are better in patients under statin treatment at the moment of stroke. Patients pretreated with statins showed better survival, less severe neurologic deficits, and improved outcomes when they were treated with thrombolysis.

However, it is unknown whether statin treatment in stroke patients is effective when it is administrated during the acute stage.

Based on strong supportive evidence in human and experimental animals which support theoretical superiority of rosuvastatin, this study will test a hypothesis that a high dose of rosuvastatin is effective in preventing recurrence during the first month after onset in ischemic stroke patients and should be given to all patients from their onset.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 20 years of age
2. Ischemic stroke patients who were undertaken MRI within 48 hrs after onset of symptoms
3. Patients underwent baseline MRI (DWI, FLAIR, GRE and MRA)
4. Ischemic stroke patients with any degree of stenosis on the relevant artery of atherothrombotic origin appearing on DWI through MRA or CTA
5. Statin-naïve (untreated with statin for the past 3 months)

Exclusion Criteria:

1. Hemorrhagic stroke/ history of symptomatic hemorrhagic stroke.
2. Presence of high-risk potential cardiac sources of embolism based on the TOAST classification or other determined etiology of stroke at the time of enrollment.
3. Known major hematologic, neoplastic, metabolic, gastrointestinal or endocrine dysfunction which, in the judgment of the Investigator, may affect the subject's ability to complete the study.
4. History of malignancy, except in subjects who have been disease-free >5 years or whose only malignancy has been basal or squamous cell skin carcinoma.
5. Life-threatening illness indicating the subject is not expected to survive for at least 2 years.
6. Secondary causes of nephrotic syndrome, and/or renal dysfunction (serum creatinine >2.0 mg/dL [177 mmol/L]) at screening.
7. Significant medical or psychological condition that, in the opinion of the Investigator, would compromise the subject's safety or successful participation in the study.
8. Unreliability as a study participant based on the Investigator's knowledge of the subject, such as drug or alcohol abuse.
9. Pregnant or lactating women or women of childbearing potential who were not protected from pregnancy by an accepted method of contraception, such as the oral contraceptive pill, an intrauterine device or surgical sterilization
10. Uncontrolled hypertension defined as either a resting diastolic blood pressure of >110 mmHg or a resting systolic blood pressure of >185 mmHg recorded at screening despite blood pressure lowering therapy.
11. Clinically significant heart disease which, in the opinion of the Principal Investigator (or designee), is likely to require coronary bypass surgery, cardiac transplantation, surgical repair and/or replacement during the course of the study.
12. Subjects who have symptoms consistent with moderate or greater severity of] congestive heart failure (CHF) (New York Heart Association [NYHA] Class III or IV), or whose most recent determination of left ventricular ejection fraction (LVEF) is <0.35.
13. Triglyceride (TG) level of greater than 500 mg/dL at screening.
14. LDL level of greater than 190 mg/dL at screening.
15. Creatine kinase (CK) >3 times the upper limit of the normal (ULN) range at screening, because of the potential of statins to cause muscle abnormalities.
16. Active liver disease or hepatic dysfunction, as determined by aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]) or bilirubin levels >3 x ULN at screening, because of the potential of statins to cause disturbances in liver function.
17. Uncontrolled primary hypothyroidism (defined as thyroid stimulating hormone [TSH] >1.5 x ULN.
18. Modified Rankin scale score 4 to 6 before stroke.
19. Participation in any investigational clinical study for drug or device within 30 days prior to study entry or expectation to participate in any other investigational clinical study for drug or device during the course of this study.
20. Patients who may need conventional angiography or intervention within 14 days after enrollment.
21. Known serious hypersensitivity reactions to HMG-CoA reductase inhibitors.
22. Use of any medication listed in the Prohibited Medications Section
23. History of myopathy.
24. Patients who has Galactose intolerance,lactose intolerance,Glucose- Galactose absorption problem.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2010-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Presence Of Newly Developed DWI Lesions | During 14 days of treatment
  The objective would be to Compare the recurrence rate of ischemic strike by comparing the PRESENCE of newly developed DWI between baseline and after 14 days of treatment.

SECONDARY OUTCOMES:
Volume Of DWI Lesions With Percent Improvement Of NIHSS Score | During 14 days of treatment
  1. Percent Improvement Based On NIHSS Score Measurements At Baseline, 5 Days And 14 Days Of Treatment.
  2. Volume Of DWI Lesions

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoe Heo, MD., Ph. D, Principal Investigator — Department of Neurology, Severance Hospital, 250 Seongsan-no,Seodaemun-gu,Seoul,120-752, Korea
Locations (27):
- South Korea (27):
  - Department of Neurology, Hallym University Sacred Heart Hospital, Anyang
  - Department of Neurology Colleage of Medicine Dong-A University, Busan
  - Department of Neurology Pusan National University Hospital, Busan
  - Department of Neurology, College of Medicine Inje University, Paik Hospital, Busan
  - Department of Neurology, Fatima hospital, Changwon
  - Department of Neurology, Samsung Changwon hospital, Changwon
  - Department of Neurology, Dongsan Medical Center, Keimyung University School of Medicine, Daegu
  - Department of Neurology, Yeungnam University School of Medicine, Daegu
  - Department of Neurology Konyang University Hospital, Daejeon
  - Department of Neurology, Chonnam National University Hospital, Gwangju
  - Department of Neurology, Chosun University Hospital, Gwangju
  - Department of Neurology, Inha University Hospital, Incheon
  - Department of Neurology, National health insurance corporation ilsan Hospital, Koyang-shi
  - Department of Neurology, Severance Hospital, Seoul
  - Department of Neurology Gangnam Severance Hospital, Seoul
  - Department of Neurology Kyung Hee University East-West Neo Medical Center, Seoul
  - Department of Neurology Seoul National University Hospital, Seoul
  - Department of Neurology St. Mary's Hospital, Catholic University, Seoul
  - Department of Neurology, Ewha Womans University Hospital, Seoul
  - Department of Neurology, Hallym University Medical Center, Seoul
  - Department of Neurology, Korean University Guro hospital, Seoul
  - Department of Neurology, Kyung Hee University, College of Medicine, Seoul
  - Department of Neurology, National Medical Center, Seoul
  - Department of Neurology, Samsung Medical Center, Seoul
  - Department of Neurology, University of Ulsan,Asan Medical Center, Seoul
  - Department of Neurology,Sanggye Paik Hospital, Inje University College of Medicine, Seoul
  - Department of Neurology, Wonju Christian Hospital, Wŏnju